CLINICAL TRIAL: NCT03746509
Title: Laryngeal Vibration as a Non-invasive Treatment for Spasmodic Dysphonia
Brief Title: Laryngeal Vibration for Spasmodic Dysphonia
Acronym: SD-VTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIN-2022-30628-2; R01DC016315 (NIH)
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Spasmodic Dysphonia
Keywords: Dystonia; Spasmodic dysphonia; Laryngeal dystonia
MeSH Terms: conditions — Dysphonia; Dystonia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-High Treatment (Experimental): Participants in the low-high treatment group will receive Laryngeal Vibration (Treatment) at 100Hz frequency once a week for a duration of 4 weeks (low intensity). Then they will switch and receive laryngeal vibration at 100Hz frequency every second day of the week (high intensity) for a duration of 4 weeks.
  Interventions: Device: Laryngeal Vibration (Treatment)
- High-Low Treatment (Experimental): Participants in the high-low treatment group will receive Laryngeal Vibration (Treatment) at 100Hz frequency every second day of the week for a duration of 4 weeks (high intensity). Then they will switch and receive laryngeal vibration at 100Hz frequency once a week for a duration of 4 weeks (low intensity).
  Interventions: Device: Laryngeal Vibration (Treatment)
- Low-High Comparator (Active Comparator): Participants in the low-high comparator group will receive Laryngeal Vibration (Comparator) at 5Hz frequency once a week for a duration of 4 weeks (low intensity). Then they will switch and receive laryngeal vibration at 5Hz frequency every second day of the week (high intensity) for a duration of 4 weeks.
  Interventions: Device: Laryngeal Vibration (Comparator)
- High-Low Comparator (Active Comparator): Participants in the high-low comparator group will receive Laryngeal Vibration (Comparator) at 5Hz frequency every second day of the week for a duration of 4 weeks (high intensity). Then they will switch and receive laryngeal vibration at 5Hz frequency once a week for a duration of 4 weeks (low intensity).
  Interventions: Device: Laryngeal Vibration (Comparator)

INTERVENTIONS:
Device: Laryngeal Vibration (Treatment) — The strength of the vibration is similar to the vibration experienced from vibrating cell phones or gaming joysticks. Vibro-tactile stimulation at the applied frequency and amplitude is not known to cause pain or tissue damage. The participant may feel a mild tingling or vibrating sensation. Preliminary testing on healthy human subjects showed that at the given vibration parameters no adverse reactions occur.
  Arms: High-Low Treatment; Low-High Treatment
Device: Laryngeal Vibration (Comparator) — The strength of the vibration is similar to the vibration experienced from vibrating cell phones or gaming joysticks. Vibro-tactile stimulation at the applied frequency and amplitude is not known to cause pain or tissue damage. The participant may feel a mild tingling or vibrating sensation. Preliminary testing on healthy human subjects showed that at the given vibration parameters no adverse reactions occur.
  Arms: High-Low Comparator; Low-High Comparator

SUMMARY:
The general aim of the research is to provide scientific evidence that vibro-tactile stimulation (VTS) represents a non-invasive form of neuromodulation that can induce measurable improvements in the speech of people with spasmodic dysphonia (SD). This research addresses a clinical need to develop alternative or auxiliary treatments for a rare voice disorder with limited treatment options. A successful completion of the proposed work will be an important step in advancing laryngeal VTS as a therapeutic intervention for improving the voice symptoms in SD. Specifically, the scientific yield by achieving the specific aims is threefold: First, it will elucidate the unknown neurophysiological mechanism behind laryngeal VTS by documenting the neural changes associated with VTS. Second, it will establish that VTS can improve voice quality in SD. Third, by documenting that laryngeal VTS yields long-term benefits on voice quality in SD patients, it would provide a solid basis for a clinical trial that needs to address open questions on optimal dosage and duration of VTS-based voice therapy, the magnitude of the therapeutic effect across adductor and abductor SD and its long term efficacy.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD) is a rare voice disorder that develops spontaneously during midlife. Patients with SD typically have a strained or choked speech and report that is takes an exhausting effort to speak. The involuntary spasms of the laryngeal musculature that give rise to these symptoms almost always occur during speech. Progression is gradual in the first year and then becomes chronic for life. The cause of spasmodic dysphonia is unknown, but SD is considered to be a form of task-specific focal dystonia (FD). More women than men are affected. Current therapeutic options are limited. SD does not respond to behavioral speech therapy. It is treated primarily with Botulinum toxin injections (Botox), which provides temporary symptom relief to some, but is not well tolerated by all SD patients. At present, there is no cure for SD.

There is convergent evidence that FD is associated with kinaesthetic deficits that are also manifest in non-dystonic musculature indicating that while the motor symptoms of dystonia are focal, the associated somatosensory deficit is general. Recent work from our group (NIH 1R21DC011841) confirmed upper limb proprioceptive deficits in SD demonstrating that an underlying somatosensory deficit is also a feature of SD. In our assessment this finding opens an avenue for a missing behavioral treatment for SD. Specifically, the investigators suggest that vibro-tactile stimulation (VTS) could be the suitable tool, given that it is known to alter afferent signals from the vibrated mechanoreceptors in muscles and skin. The approach seeks to show that VTS represents a non-invasive form of neuromodulation that induces measurable improvements in the speech of SD patients. Given that SD, like other FDs, is associated with abnormally increased cortical excitation and heightened levels of neuronal synchronization, the investigators put forward that VTS can reduce sensorimotor cortical excitation in SD by desynchronizing motor cortical neuron activity as has been shown in cervical dystonia. Technically, newly available light-weight, wearable low-voltage vibrators offer, for the first time, the possibility to apply laryngeal VTS outside a controlled laboratory environment, which would be imperative for the technology to be clinically useful. In general, one needs to demonstrate that a) VTS induces measurable improvements in voice quality, b) that it induces measurable changes in somatosensory and motor cortical activation that would provide insight into the underlying neural mechanism of its potential effectiveness. Thus, the proposal has the following specific aims:

1. Demonstrate that a one-time, prolonged application of VTS produces acute improvements in SD voice quality that are retained up to 60 minutes past cessation of VTS. A pre- and post-training comparison showing significant voice improvements in the SD group as measured by self-report (Effort Scale), clinical assessment (Consensus Auditory-Perceptual Evaluation of Voice - CAPE-V), as the reduction in the number of voice breaks and determining cepstral peak prominence will realize this goal. The investigators' preliminary data show that VTS induces improvements in voice quality in SD patients as measured by these markers.
2. Demonstrate that repeated prolonged VTS produces long lasting improvements in SD voice quality that are retained for up to 3 months. SD patients will participate in an 8-week in-home VTS training program. After randomization to either a treatment or sham group (ineffective low frequency VTS), patients will start in low or high intensity training group (1 vs. 3 sessions/wk) and cross-over after 4 weeks. Showing that significant long-term voice improvements in the VTS treatment group as assessed by objective measures of voice/speech production (see aim 1) will persist over a period of 11 weeks will realize this goal.
3. Demonstrate that the application of VTS induces acute desynchronization of cortical activity in SD, which would provide neurophysiological evidence on the assumed effectiveness of VTS. Verifying that VTS is associated with short-latency characteristic changes in somatosensory and motor cortical processing as measured by electroencephalography (EEG) and documenting that these changes indicate decreased alpha and beta-band activity in sensorimotor cortical areas will achieve this goal. The investigators' preliminary data show that VTS suppresses low frequency neural activity at the somatosensory and motor cortices in healthy and SD participants. Obtaining longitudinal EEG data during VTS training (aim 2), will allow the investigators to monitor long-term changes in cortical activation due to laryngeal VTS and to associate them with changes in voice quality.

Impact. This is the first systematic study on the effect of VTS on SD voice symptoms. The proposal aligns with PA-14-236 (Advancing Research in Voice Disorders) with its emphasis on understanding voice disorders and improving diagnosis and treatment. If successful, the work of the proposal would lay the scientific foundation for a clinical trial to examine the usefulness of the approach in a larger patient sample. It would document the sensorimotor cortical activation patterns associated with SD and the longitudinal changes in cortical responses to VTS. It would promote development of wearable, user-programmable medical devices that could apply VTS while monitoring its effect on voice production in real-time. Ultimately, VTS would enlarge the available therapeutic arsenal by either augmenting existing Botox therapy or becoming an alternative intervention option for patients who do not tolerate Botox injections.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of adductor SD for a minimum of 6 months with documented symptom relief after botox injection

Exclusion Criteria:

* abductor SD
* patients with other voice disorders such as muscle tension dysphonia that share some of the symptomology with SD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Konczak, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khosravani S, Mahnan A, Yeh IL, Aman JE, Watson PJ, Zhang Y, Goding G, Konczak J. Laryngeal vibration as a non-invasive neuromodulation therapy for spasmodic dysphonia. Sci Rep. 2019 Nov 29;9(1):17955. doi: 10.1038/s41598-019-54396-4. PMID 31784618
- [Result] Konczak J, Bhaskaran D, Elangovan N, Oh J, Goding GS, Watson PJ. Effects of an 11-week vibro-tactile stimulation treatment on voice symptoms in laryngeal dystonia. Front Neurol. 2024 May 30;15:1403050. doi: 10.3389/fneur.2024.1403050. eCollection 2024. PMID 38872829
- See also: Invesitgator laboratory website summarizing study results — https://hsc.umn.edu/vibro-tactile-stimulation-topic/laryngeal-vibration-treatment-voice-disorder

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Fairview Voice Clinic at the University of Minnesota and through e-mail advertisements sent by the National Spasmodic Dysphonia Association as well as social media platforms.
  Recruitment began in the Fall of 2018.
Period: Overall Study
Arm/Group | Low-High Treatment | High-Low Treatment | Low-High Comparator | High-Low Comparator
Started | 11 | 10 | 11 | 10
Completed | 7 | 8 | 9 | 9
Not Completed | 4 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-High Treatment | High-Low Treatment | Low-High Comparator | High-Low Comparator | Total
Number analyzed (Participants) | 11 | 10 | 11 | 10 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 8 | 20
  >=65 years | 7 | 6 | 7 | 2 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 7 | 4 | 23
  Male | 4 | 5 | 4 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 11 | 10 | 10 | 8 | 39
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Voice Assessment During First Visit
Description: Smoothed Cepstral Peak Prominence (CPPS) is an indicator of voice quality. It is measured in decibels. CPPS was measured from the voice signals of each participant during each study visit, and relative CPPS was calculated before and after vibration was applied on the laryngeal muscles of the participants. An increase in CPPS value indicates an improvement in voice symptoms.
Time Frame: Testing performed in lab at Week 1
Measure: Median (Inter-Quartile Range); unit: decibel
Arm/Group | Low-High Treatment | High-Low Treatment | Low-High Comparator | High-Low Comparator
Number analyzed (Participants) | 10 | 10 | 10 | 9
decibel | 0.045 [-0.79 to 1.28] | 0.17 [-0.91 to 1.05] | 0.13 [0.01 to 1.14] | -0.47 [-0.64 to 0.56]

2. Primary Outcome: Final Voice Assessment
Description: Smoothed Cepstral Peak Prominence (CPPS) which is an indicator of voice quality was measured in participants. CPPS was measured in participants during the first visit, and relative CPPS was calculated before and after vibration was applied on the laryngeal muscles of the participants.
Time Frame: Testing performed in lab at week 11
Measure: Median (Inter-Quartile Range); unit: decibel
Arm/Group | Low-High Treatment | High-Low Treatment | Low-High Comparator | High-Low Comparator
Number analyzed (Participants) | 8 | 10 | 7 | 8
decibel | 0.96 [0.71 to 1.30] | 0.55 [-0.82 to 0.63] | 0.64 [0.21 to 1.37] | 0.23 [-0.01 to 0.38]

3. Secondary Outcome: Measuring of Cortical Activity Using Electroencephalography (EEG) (Baseline)
Description: Cortical activity before, during, and after the vibration will be recorded via a a 64-channel EEG system at a sampling frequency of 512 Hz.
Time Frame: Testing performed in lab at Week 1
Reporting Status: Not Posted

4. Secondary Outcome: Final Measuring of Cortical Activity Using Electroencephalography (EEG) to Measure Change From Baseline
Description: as for outcome 3
Time Frame: Testing performed in lab at Week 11
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | Low-High Treatment | High-Low Treatment | Low-High Comparator | High-Low Comparator
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Dosage was limited to apply vibro-tactile stimulation for one day or days per week for 20 min/day. It is unclear how a more frequent or longer application of the stimulation will affect voice outcome in people with laryngeal dystonia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03746509/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03746509/ICF_001.pdf